CLINICAL TRIAL: NCT02139020
Title: Prospective Collection of Plasma Samples From Patients Treated With Molecular Targeted Therapies for Squamous Cell Carcinoma of the Head and Neck
Brief Title: Collection of Plasma Samples for Squamous Cell Carcinoma of the Head and Neck Patients
Status: Recruiting | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: UCL-ONCO 2013-01
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Targeted therapies; Plasma samples
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One EDTA tube is collected at the beginning of the study and there are only plasma samples at baseline, during treatment, and at progression.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Patients with squamous cell carcinoma of the head and neck, targeted therapies, plasma samples:
  * Group 1 = patients treated with radiation therapy and cetuximab according to Bonner et al [11]
  * Group 2 = patients treated with cetuximab in combination with chemotherapy according to Vermorken et al. [10]
  * Group 3 = patients treated with a molecular targeted agent as a part of a clinical study
  Interventions: Other: Plasma samples

INTERVENTIONS:
Other: Plasma samples — Plasma samples at baseline (and one whole blood sample) and at every radiological evaluations

SUMMARY:
The investigators will collect plasma samples at baseline, during treatment, and at progression.

DETAILED DESCRIPTION:
In this study, the investigators will collect plasma samples at baseline, during treatment, and at progression. This plasma bank will be used to study the potential value of some biomarkers to predict treatment activity or resistance to cetuximab or other targeted agents

ELIGIBILITY:
Inclusion Criteria:

* patients treated with radiation therapy and cetuximab according to Bonner et al
* patients treated with cetuximab in combination with chemotherapy according to Vermorken et al.
* patients treated with a molecular targeted agent as a part of a clinical study

Exclusion Criteria:

* patients with another type of head and neck cancer
* patients non treated with targeted therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PATIENTS TREATED WITH MOLECULAR TARGETED THERAPIES FOR SQUAMOUS CELL CARCINOMA OF THE HEAD AND NECK
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-02; Primary Completion 2033-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Prospective storage of plasma samples of patients treated with cetuximab or other targeted agents | one year after the collection
  All the analyses will be done when we have enough of collected samples

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal Machiels, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (5):
- Belgium (5):
  - Clinique Saint-Pierre, Ottignies, Brabant Wallon
  - Grand Hôpital de Charleroi, Charleroi, Hainaut
  - Centre Hospitalier Jolimont-Lobbes-Nivelles-Tubize, Haine-Saint-Paul
  - CHU Liège, Liège
  - Clinique et Maternité Sainte-Elisabeth, Namur